CLINICAL TRIAL: NCT00005743
Title: Exercise Adherence in a Behavioral Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized
Other Study IDs: 4967; R29HL056127 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise
Behavioral: weight loss

SUMMARY:
To develop intervention strategies that improve long-term exercise adherence in obese adults in in order to improve long-term weight loss.

DETAILED DESCRIPTION:
BACKGROUND:

Even though exercise improves long-term weight loss maintenance and reduces the risks of cardiovascular disease and Type II diabetes mellitus, obese adults are prone to drop out of exercise programs. Dr. Jakicic's prior findings suggest that exercise adherence can be enhanced and short-term weight loss can be improved by making exercise more convenient via prescribing exercise in multiple short bouts, rather than one bout per day. Effects on long-term exercise adherence and weight loss have not been examined, however. His findings also suggest that providing more exercise options by placing exercise equipment in the home may also increase adherence, as evidenced by a significant correlation between the presence of home exercise equipment and physical activity. However, no experimental studies have tested whether placing exercise equipment in the home actually increases exercise adherence and weight loss.

DESIGN NARRATIVE:

The study tested the hypothesis that prescribing exercise in multiple short bouts would improve long-term exercise adherence and long-term weight loss, and that the addition of home exercise equipment would further improve these outcomes. A total of 148 overweight women were recruited and randomized to one of three treatments: 1) long-bout exercise; 2) short-bout exercise; 3) short- bout exercise + home exercise equipment. All subjects participated in an 18-month behavioral weight loss program, in which body weight was assessed at 0, 6, 12, and 18 months and exercise adherence was assessed throughout the 18 months. Cardiorespiratory fitness and cardiovascular disease risk factors were measured at 0, 6, and 18 months.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-05; Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Jakicic — The Miriam Hospital

REFERENCES:
- [Background] Jakicic JM, Winters C, Lang W, Wing RR. Effects of intermittent exercise and use of home exercise equipment on adherence, weight loss, and fitness in overweight women: a randomized trial. JAMA. 1999 Oct 27;282(16):1554-60. doi: 10.1001/jama.282.16.1554. PMID 10546695
- [Background] Jakicic JM, Winters C, Lagally K, Ho J, Robertson RJ, Wing RR. The accuracy of the TriTrac-R3D accelerometer to estimate energy expenditure. Med Sci Sports Exerc. 1999 May;31(5):747-54. doi: 10.1097/00005768-199905000-00020. PMID 10331898
- [Background] Dunn AL, Andersen RE, Jakicic JM. Lifestyle physical activity interventions. History, short- and long-term effects, and recommendations. Am J Prev Med. 1998 Nov;15(4):398-412. doi: 10.1016/s0749-3797(98)00084-1. PMID 9838980
- [Background] Jakicic JM, Lang W, Wing RR. Do African-American and Caucasian overweight women differ in oxygen consumption during fixed periods of exercise? Int J Obes Relat Metab Disord. 2001 Jul;25(7):949-53. doi: 10.1038/sj.ijo.0801632. PMID 11443491
- [Background] Jakicic JM, Wing RR, Winters-Hart C. Relationship of physical activity to eating behaviors and weight loss in women. Med Sci Sports Exerc. 2002 Oct;34(10):1653-9. doi: 10.1097/00005768-200210000-00018. PMID 12370568
- [Background] Gallagher KI, Jakicic JM, Kiel DP, Page ML, Ferguson ES, Marcus BH. Impact of weight-cycling history on bone density in obese women. Obes Res. 2002 Sep;10(9):896-902. doi: 10.1038/oby.2002.123. PMID 12226138